CLINICAL TRIAL: NCT02526446
Title: A Randomized, Wait-list Controlled Trial of Self-administered Acupressure for Symptom Management Among Chinese Family Caregivers With Caregiver Stress
Brief Title: Self-administered Acupressure for Symptom Management of Caregiver Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Agnes Tiwari, Professor and Head of School of Nursing, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW 15-367
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Stress
Keywords: Chinese; caregiver stress; self-administered acupressure
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-administered acupressure (Experimental): The intervention consists of a total of 28 hours over a period of 8 weeks. It comprises of individual learning and practice, self-practice at home, and home follow-up.
  Interventions: Behavioral: Self-administered acupressure
- Wait-list control (Other): The control group will receive a wait-list control condition (the same self-administered acupressure intervention but after the intervention group has completed the treatment condition).
  Interventions: Other: wait-list control

INTERVENTIONS:
Behavioral: Self-administered acupressure — The intervention consists of a total of 28 hours over a period of 8 weeks:
  i) Individual learning and practice: The training session will be one-on-one provided twice a week for two consecutive weeks (5 hours) in the participant's home.
  ii) Self-practice at home: From 3rd to 8th week, participant will engage in self-administered acupressure at home for 15 minutes twice a day for 6 weeks (21 hours).
  iii) Home follow-up: During the 3rd and 4th week (i.e. after the 2-week training session), a 1-hour home visit will be conducted for reinforcement of learning and self-practice by the same team of trainers once a week for 2 weeks (2 hours).
  Arms: Self-administered acupressure
Other: wait-list control — The control group will receive a wait-list control condition (the same self-administered acupressure intervention but after the intervention group has completed the treatment condition).
  Arms: Wait-list control

SUMMARY:
This proposed study is to evaluate the effectiveness of a self-administered acupressure intervention on caregiver stress and associated distress symptoms of fatigue, insomnia and depression in Chinese family caregivers of an elderly family member.

DETAILED DESCRIPTION:
Taking care of an elderly family member can be stressful and family caregivers are at risk for emotional, mental and physical health problems arising from caregiver stress. Although a variety of psychosocial and pharmacological strategies have been developed to reduce caregiver stress, the efficacy in mitigating caregiver distress is modest. Acupressure, a non-invasive technique of Traditional Chinese Medicine (TCM) by applying pressure on acupoints, has been successfully used for management of multiple symptoms without adverse effects. Thus, this study using a randomized, wait-list controlled trial is to evaluate the effectiveness of self-administered acupressure intervention on caregiver stress and associated distress symptoms of fatigue, insomnia or depression. A total of 200 Chinese family caregivers with caregiver stress and stress related symptoms of fatigue, insomnia or depression will be recruited from a community setting in Hong Kong and randomized to receive either a self-administered acupressure intervention or wait-list condition. The self-administered acupressure intervention will comprise (i) 5-hr individual learning and training session in the first 2 weeks, (ii) 2-hr home-visit reinforcement during 3rd and 4th week, and (iii) a total of 21-hr self-practice at home over 6 weeks. It is hypothesized that the family caregivers in the intervention group will have, upon completion of the program, lower levels of caregiver stress, lower scores of fatigue, insomnia, and depression with improved health-related quality of life as compared with that in the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Chinese woman or man, 21 years of age or older, able to communicate in Cantonese or Putonghua,
* Primary caregiver of an elderly family member aged ≥ 65 years,
* Providing unpaid care to the care recipient at no less than 14 hours per week,
* Primarily responsible for making day-to-day decisions and providing assistance to the care recipient in tasks relating to activities of daily living (e.g. bathing, dressing, toileting etc.) and/or instrumental activities of daily living (e.g. housework, grocery shopping, preparing meals, managing medications etc.), and
* Screened positive for caregiver stress (a summed score of ≥ 25 as measured by the Caregiver Burden Inventory), with symptoms of fatigue (a mean score of ≥ 4 as measured by the Piper Fatigue Scale), insomnia (a global score of > 5 as measured by the Pittsburgh Sleep Quality Index), OR depression (a total score of ≥ 10 as measured by the Patient Health

Exclusion Criteria:

* Cognitive impairment (a Mini Mental State Examination (MMSE) score of ≤ 23), or
* Major chronic illness (e.g. cancer) or currently taking any medications (e.g. opiates) that may prevent them from performing the intervention, or
* Participated in intervention studies involving acupressure or acupuncture previously.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in caregiver stress | Baseline (T0, on entry to study before intervention), (ii) post-training (T1, 2-week later on completion of the group training, (iii) post-intervention (T2, 6-week later on completion intervention, and (iv) follow-up (T3, 4-week post-intervention)
  Score on measure of caregiver stress by Chinese version of the Caregiver Burden Inventory (C-CBI)

SECONDARY OUTCOMES:
Fatigue score | Baseline (T0, on entry to study before intervention), (ii) post-training (T1, 2-week later on completion of the group training, (iii) post-intervention (T2, 6-week later on completion intervention, and (iv) follow-up (T3, 4-week post-intervention)
  Score on measure of Fatigue by Chinese Piper Fatigue Scale (C-PFS)
Insomnia score | Baseline (T0, on entry to study before intervention), (ii) post-training (T1, 2-week later on completion of the group training, (iii) post-intervention (T2, 6-week later on completion intervention, and (iv) follow-up (T3, 4-week post-intervention)
  Score on measure of Insomnia by Chinese Pittsburgh Sleep Quality Index (C-PSQI)
Depression score | Baseline (T0, on entry to study before intervention), (ii) post-training (T1, 2-week later on completion of the group training, (iii) post-intervention (T2, 6-week later on completion intervention, and (iv) follow-up (T3, 4-week post-intervention)
  Score on measure of Depression by Chinese Patient Health Questionnaire (C-PHQ);
Caregiver's quality of life (QoL) | Baseline (T0, on entry to study before intervention), (ii) post-training (T1, 2-week later on completion of the group training, (iii) post-intervention (T2, 6-week later on completion intervention, and (iv) follow-up (T3, 4-week post-intervention)
  Score on measure of Quality of Life by Chinese SF-12 version 2 Health Survey (SF-12v2)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Tiwari, PhD, Principal Investigator — School of Nursing, HKU
Locations (1):
- HKSKH Lady MacLehose Center, Hong Kong, Hong Kong

REFERENCES:
- [Result] Tiwari A, Fong DY, Yuen KH, Yuk H, Pang P, Humphreys J, Bullock L. Effect of an advocacy intervention on mental health in Chinese women survivors of intimate partner violence: a randomized controlled trial. JAMA. 2010 Aug 4;304(5):536-43. doi: 10.1001/jama.2010.1052. PMID 20682933
- [Result] Zhang Y, Shen CL, Peck K, Brismee JM, Doctolero S, Lo DF, Lim Y, Lao L. Training Self-Administered Acupressure Exercise among Postmenopausal Women with Osteoarthritic Knee Pain: A Feasibility Study and Lessons Learned. Evid Based Complement Alternat Med. 2012;2012:570431. doi: 10.1155/2012/570431. Epub 2012 Oct 23. PMID 23193423
- [Result] Tiwari A, Chan CL, Ho RT, Tsao GS, Deng W, Hong AW, Fong DY, Fung HY, Pang EP, Cheung DS, Ma JL. Effect of a qigong intervention program on telomerase activity and psychological stress in abused Chinese women: a randomized, wait-list controlled trial. BMC Complement Altern Med. 2014 Aug 15;14:300. doi: 10.1186/1472-6882-14-300. PMID 25127878
- [Result] Yeung WF, Chung KF, Poon MM, Ho FY, Zhang SP, Zhang ZJ, Ziea ET, Wong VT. Acupressure, reflexology, and auricular acupressure for insomnia: a systematic review of randomized controlled trials. Sleep Med. 2012 Sep;13(8):971-84. doi: 10.1016/j.sleep.2012.06.003. Epub 2012 Jul 25. PMID 22841034
- [Result] Wang XM, Walitt B, Saligan L, Tiwari AF, Cheung CW, Zhang ZJ. Chemobrain: a critical review and causal hypothesis of link between cytokines and epigenetic reprogramming associated with chemotherapy. Cytokine. 2015 Mar;72(1):86-96. doi: 10.1016/j.cyto.2014.12.006. Epub 2015 Jan 5. PMID 25573802
- [Derived] Cheung DST, Tiwari A, Yeung WF, Yu DSF, So MKP, Chau PH, Wang XM, Lum TYS, Yuk Fung HYK, Ng BYM, Zhang ZJ, Lao L. Self-Administered Acupressure for Caregivers of Older Family Members: A Randomized Controlled Trial. J Am Geriatr Soc. 2020 Jun;68(6):1193-1201. doi: 10.1111/jgs.16357. Epub 2020 Feb 25. PMID 32096884
- [Derived] Tiwari A, Lao L, Wang AX, Cheung DS, So MK, Yu DS, Lum TY, Yuk Fung HY, Yeung JW, Zhang ZJ. Self-administered acupressure for symptom management among Chinese family caregivers with caregiver stress: a randomized, wait-list controlled trial. BMC Complement Altern Med. 2016 Oct 28;16(1):424. doi: 10.1186/s12906-016-1409-1. PMID 27793197